CLINICAL TRIAL: NCT03238794
Title: Effect of Weight Loss Through RYGB Versus Weight Loss Through Caloric Restriction on the Bile Acid Pathway
Brief Title: Bariatric Surgery Versus Diet Alone in the Bile Acid Pathway and Weight Loss
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Andres J. Acosta, M.D., Ph.D., Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 16-008664; K23DK114460 (NIH)
Record Dates: First submitted 2017-08-01; First posted 2017-08-03 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Obesity
Keywords: Body Mass Index; gastric; bypass; bariatric surgery; bile acid; weight loss; diet; low calorie
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Gastric Bypass; Caloric Restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Roux-En-Y Gastric Bypass (RYGB) (Active Comparator): Participants will have elected to have RYGB surgery per standard of care.
  Interventions: Procedure: Roux-En-Y Gastric Bypass
- Low-calorie Diet (Active Comparator): Participants will have a low-calorie diet prescribed by a registered dietitian.
  Interventions: Other: Low-calorie Diet

INTERVENTIONS:
Procedure: Roux-En-Y Gastric Bypass — Food will be consumed as directed by their doctor as standard of care. A food log will be completed the week before visits 3 and 5.
  Other Names: RYGB
  Arms: Roux-En-Y Gastric Bypass (RYGB)
Other: Low-calorie Diet — Food will be consumed as Week one will be liquid 400 to 500 kcal/day, weeks 2,3, and 4 will consist of 500-600 kcal/day of pureed food, weeks 5-8 will consist of 600-800 kcal/day of mechanical-soft food, weeks 9-12 will consist of 800 to 1000 kcal/day of soft foods, and the remainder of the study participants will be given 1000 to 1200 kcal/day of regular food.
  Arms: Low-calorie Diet

SUMMARY:
It is unknown whether the bile acid pathway reacts differently to weight loss resulting from Roux-En-Y Gastric Bypass (RYGB) surgery than weight loss resulting from caloric restriction alone.

DETAILED DESCRIPTION:
Participants will be placed into two groups. The Roux-En-Y Gastric Bypass (RYGB) group will consist of participants who will have elected to have RYGB at the Mayo Clinic Bariatric Center of Excellence. The Diet group will have a low-calorie diet prescribed by a registered dietitian. Both groups will collect stool from every bowel movement 2 days before presenting for baseline testing. Both group participants will present for baseline testing after an overnight fast and before intervention (RYGB or low calorie diet). Participants will consume a standard breakfast provided by study staff and blood samples will be collected at -15, 0, 15, 30,45,60,90,120,150,180,210,240,300,360 minutes. Appetite and satiation ratings will be recorded via questionnaires during that day every 15 minutes for the first 90 minutes, then every 30 minutes. Participants will repeat this regimen again after losing 7% of their body weight after having RYGB or low calorie diet.

ELIGIBILITY:
Inclusion Criteria:

* Women of childbearing potential will have negative pregnancy tests within 48 hours of enrolment.
* BMI: ≥ 40
* Individuals who have elected to have RYGB at the Mayo Clinic Bariatric Center of Excellence, and individuals with a BMI ≥40 who are otherwise healthy with controlled cardiac, pulmonary, gastrointestinal, hepatic, renal, hematological, neurological, or endocrine disorders. The RYGB participants will be invited to participate when their surgery is scheduled at the Mayo Clinic Bariatric Center of Excellence.
* The non-RYGB participants (BMI ≥40) will be otherwise healthy individuals with no unstable psychiatric disease and no unstable cardiac, pulmonary, gastrointestinal, hepatic, renal, hematological, neurological, or endocrine disorders.

Exclusion Criteria:

* History of abdominal surgery including cholecystectomy and other than appendectomy, Caesarian section or tubal ligation.
* Positive history of chronic gastrointestinal diseases, or systemic disease that could affect gastrointestinal motility, or use of medications that may alter gastrointestinal motility, appetite or absorption, e.g., orlistat, phentermine.
* Significant untreated psychiatric dysfunction based upon screening with the Hospital Anxiety and Depression Inventory (HAD), a self-administered alcoholism screening test (AUDIT-C) and the Questionnaire on Eating and Weight Patterns (binge eating disorders and bulimia). If such a dysfunction is identified by a depression or anxiety score >11 or difficulties with substance or eating disorders, the participant will be excluded and given a referral letter to his/her primary care doctor for further appraisal and follow-up. The AUDIT-C is a 3-item alcohol screening questionnaire that reliably identifies participants who are hazardous alcohol drinkers or have active alcohol use disorders. In men, a score of 4 or more is above the recommended limits will be reviewed by study personnel. In women, a score of 3 or more is above the recommended limits will be reviewed by study personnel. However when the points are above recommended limits, the provider will review the patient's alcohol intake over the past few months to confirm accuracy and determine study eligibility.
* Any acute or chronic condition or other disease that, in the opinion of the Investigator, would limit the subject's ability to complete and/or participate in this clinical study.Participant activities:
* If recruited for the investigation participants will be asked to refrain from donating blood; refrain from participating in other research studies; avoid taking any additional over the counter or prescription medications or herbal supplements that have not been reviewed and approved by the physician or the study coordinator until the study has been completed

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-05-17 (Actual); Primary Completion 2027-01-11 (Estimated); Study Completion 2027-01-11 (Estimated)

PRIMARY OUTCOMES:
Change in Bile Acid (BA) excretion | baseline, 12 weeks
  Total Fecal BA excretion change measured in mcmoles/48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Andres J Acosta, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials